CLINICAL TRIAL: NCT07281222
Title: Evaluation of the FYNA Research OPM MEG Device for Locating Epileptic Foci as Part of Pre-surgical Assessment of Epilepsy
Acronym: EPI-OPM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: MAG4Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL24_0886; 2025-A02262-47 (Other: ID-RCB)
Record Dates: First submitted 2025-11-20; First posted 2025-12-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy
Keywords: Epilepsy; magnetoencephalography; MEG; Fyna Research; epilepsy surgery; epileptic foci
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug-resistant epilepsy patients who are candidates for epilepsy surgery (Experimental): Patients are drug-resistant epilepsy who are candidates for whom the following are decided and planned:
  either 1) a surgical procedure to resect the epileptogenic zone without prior intracranial EEG recording or 2) intracranial EEG recording necessary prior to a possible cortical resection procedure They will undergo two imaging examinations specific to the study: OPM MEG examination with the FYNA Research device evaluated in this study and a conventional SQUID MEG examination. If necessary (not already performed/available), the will undergo a brain MRI during a single visit.
  Interventions: Device: MEG OPM; Device: MEG SQUID

INTERVENTIONS:
Device: MEG OPM — The OPM MEG sensor (FYNA Research device) is a new sensor technology for MEG (magnetoencephalography). It consists of 48 detectors (helium-4 magnetometers) that are positioned on the patient's head using a support system that can be adjusted to fit the size of their head. The patient goes to the MEG center at CERMEP (patients included in Lyon) or INS (patients included in Marseille), changes clothes, and removes any makeup. Metal-free clothing designed for MEG is provided. The tracking coils are put in place. The patient is then placed in the MEG, and their positioning and comfort are checked again.
  The OPM MEG acquisition takes about 60 minutes.
Device: MEG SQUID — The MEG SQUID is the classical MEG (magnetoencephalography). It consists of a set of sensors placed in a rigid helmet, in contact with the head. The patient goes to the MEG center at CERMEP (patients included in Lyon) or INS (patients included in Marseille), changes clothes, and removes any makeup. Metal-free clothing designed for MEG is provided. The tracking coils are put in place. The patient is then placed in the MEG, and their positioning and comfort are checked again.
  The OPM MEG acquisition takes about 60 minutes.

SUMMARY:
The success of epilepsy surgery depends largely on the reliability of the preoperative localization of the epileptogenic zone. The conventional method for determining the area to be removed is based on a complex assessment involving an electroencephalogram (EEG) coupled with simultaneous video recording of seizures (video SEEG), a brain MRI, and a fluorodeoxyglucose positron emission tomography scan (PET-FDG).

At present, epilepsy surgery cannot cure all patients. Since the prognosis for surgery depends primarily on the ability to delineate the epileptogenic zone, it is essential to develop new diagnostic approaches that can accurately detect epileptic foci.

MEG (magnetoencephalography) is a non-invasive brain mapping technique based on the magnetic fields created by neuronal activity. Numerous studies have shown that it is a highly effective technique for locating epileptic foci, and more accurate than EEG. However, MEG remains relatively uncommon (three centers in France) because current conventional systems (MEG SQUID) are difficult to use, expensive, require significant structural constraints for installation, and are not very sensitive (sensors are distant from the scalp).

Mag4Health has developed a new MEG device, the "MEG FYNA Research", which records brain magnetic activity using 48 or 96 sensors (4He optical pumping magnetometers, or "OPMs"). Compared to conventional MEG (SQUID MEG), this OPM MEG technology is more compact, less expensive, more sensitive, and allows the sensors to be placed directly on the scalp.

The EPI-OPM study is a prospective, uncontrolled, bicenter clinical investigation that aims to evaluate the diagnostic performance of this device.

The main objective is to assess the value of the OPM MEG device for localizing the epileptogenic zone compared to the reference method in epileptic patients undergoing epilepsy surgery.

Patients (children and adults) will be enrolled at the Lyon University Hospital and the Marseille University Hospital.

Each patient will undergo an OPM MEG examination and a SQUID MEG examination (SQUID MEG only for patients in Lyon), in addition to the clinical procedures performed as part of routine care: intracranial EEG recording (SEEG) and MRI if necessary, followed by surgery to resect the epileptic focus.

The performance of the OPM MEG device in locating epileptic foci will be validated by surgical results and invasive EEG recordings. The localization of epileptic foci using the OPM MEG system will be compared with that obtained using the SQUID MEG system (conventional MEG) and other pre-surgical assessment tests carried out as part of routine care. Finally, we will describe tolerance to the recordings and assess overall comfort and feasibility using appropriate questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 6 to 65
2. Patients suffering from partial epilepsy that has been developing for at least 2 years, drug-resistant, regardless of the presumed topographical origin or suggested cause (lesional with or without MRI abnormality) and for whom the following have been decided and planned:

   either i) a surgical procedure to resect the epileptogenic zone without prior intracranial EEG recording or ii) intracranial EEG recording necessary before a possible cortical resection procedure
3. Patients who have undergone routine prolonged scalp video EEG recording showing interictal paroxysmal abnormalities
4. Patients motivated to participate effectively in the project
5. Patients who have signed an informed consent form to participate in the study

Exclusion Criteria:

1. Patients with neurological or psychiatric disorders or a history of neurological or psychiatric disorders, sleep disorders other than epilepsy that may impact the variability or quality of the data or the cooperation and retention of the participant, which will be assessed by the principal investigator or co-investigator during the inclusion interview.
2. Patients with contraindications common to MEG and MRI examinations:

   * Metal in the body that is incompatible with the examination (pacemaker, implanted pump including insulin pump, neurostimulator, cochlear implants or other hearing devices, metal prosthesis, intracerebral/surgical clips for aneurysms, implantable defibrillators, ferromagnetic foreign bodies in the eyes or brain in the upper body, ventriculoperitoneal neurosurgical shunt valves, dental braces or steel pivots for dental root canals, ferromagnetic foreign bodies in the upper body)
   * Claustrophobia
3. Pregnant women, breastfeeding women, or women who have given birth within the last 6 months.
4. Patients under guardianship, curatorship, or judicial protection
5. Patients deprived of their liberty
6. Patients not affiliated with a social security system or beneficiaries of such a system

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of cases in which the location of epileptic foci identified by MEG OPM confirmed the location identified by pre-surgical assessment (EEG, SEEG, MRI, PET-FDG) when surgery was successful, one year after its completion (composite outcome) | 1 year after surgery (18 months after inclusion)
  To do this, the existence of a spatial overlap between the location of the epileptic focus in MEG and the area operated on in patients will be assessed.
  The location of the area operated on in cured patients is considered to be the reference location of the epileptogenic zone.
  For each patient included, the location of the preoperative MEG epileptic focus will be determined by source modeling applied to the detected epileptic spikes.
  The area operated on will be determined on the postoperative MRI, and the success of the operation will be determined by the Engel score, which summarizes the postoperative evolution of epilepsy in terms of seizure frequency in the context of routine care.

SECONDARY OUTCOMES:
Percentage of cases in which the location of epileptic foci identified by MEG OPM differs from the location identified by conventional pre-surgical assessment (EEG, SEEG, MRI) when surgery was unsuccessful, 1 year after surgery. | 1 year after surgery (18 months after inclusion)
  To do this, the existence of a spatial overlap between the location of the epileptic focus in MEG and the area operated on in patients will be assessed.
  The location of the area operated on in cured patients is considered to be the reference location of the epileptogenic zone.
  For each patient included, the location of the preoperative MEG epileptic focus will be determined by source modeling applied to the detected epileptic spikes.
  The area operated on will be determined on the postoperative MRI, and the success of the operation will be determined by the Engel score, which summarizes the postoperative evolution of epilepsy in terms of seizure frequency in the context of routine care.
Percentage of congruence between the location of the epileptic focus determined by OPM MEG source modeling and the area of seizure onset estimated by SEEG. | 3 months after inclusion (Day of the SEEG Exploration)
  For each patient included, the location of the MEG OPM epileptic focus will be determined by source modeling applied to the detected epileptic spikes.
  The seizure onset zone in SEEG will be determined by analyzing the SEEG signals obtained as part of routine care.
  For each patient, the spatial overlap between the area modeled in MEG and the seizure onset zone in SEEG will be determined, allowing good or poor congruence to be determined.
Percentage of congruence between the location of the epileptic focus determined by OPM MEG source modeling and the location of the epileptic focus determined by SQUID MEG source modeling. | Day of the MEG visit (day of inclusion)
  For each patient included, the location of the epileptic focus will be determined using OPM MEG and SQUID MEG source modeling applied to the detected epileptic spikes.
  For each patient, the spatial overlap between the area modeled using OPM MEG and the area modeled using SQUID MEG will be determined, allowing good or poor congruence to be identified.
Percentage of cases in which the location of epileptic foci identified by MEG SQUID confirmed the location identified by conventional pre-surgical assessment (EEG, SEEG, MRI) when surgery was successful, one year after its completion. | 1 year after surgery (18 months after inclusion)
  To do this, the existence of a spatial overlap between the location of the epileptic focus in MEG SQUID and the area operated on in patients will be evaluated.
  The location of the area operated on in cured patients is considered to be the reference location of the epileptogenic zone.
  For each patient included, the location of the epileptic focus by MEG SQUID will be determined by source modeling applied to the detected epileptic spikes.
  The area operated on will be determined on the postoperative MRI, and the success of the operation will be determined by the Engel score, which summarizes the postoperative evolution of epilepsy in terms of seizure frequency in the context of routine care.
Percentage of cases in which the location of epileptic foci identified by MEG SQUID confirmed the location identified by conventional pre-surgical assessment (EEG, SEEG, MRI, PET-FDG) when surgery was successful, one year after its completion. | 1 year after surgery (18 months after inclusion)
  To do this, the existence of a spatial overlap between the location of the epileptic focus in MEG SQUID and the area operated on in patients will be assessed.
  The location of the area operated on in cured patients is considered to be the reference location of the epileptogenic zone.
  For each patient included, the location of the epileptic focus by MEG SQUID will be determined by source modeling applied to the detected epileptic spikes.
  The area operated on will be determined on the postoperative MRI, and the success of the operation will be determined by the Engel score, which summarizes the postoperative evolution of epilepsy in terms of seizure frequency in the context of routine care.
Percentage of congruence between the area modeled in MEG OPM and the area of seizure onset estimated in MEG SQUID | Day of the MEG visit (Day of inclusion)
  For each patient included, the location of the epileptic focus MEG (OPM and SQUID) will be determined by source modeling applied to the detected epileptic spikes.
  For each patient, the spatial overlap between the area modeled in MEG OPM and the area modeled in MEG SQUID will be determined, allowing good or poor congruence to be determined.
Percentage of congruence between the location of the epileptogenic zone determined by MRI and the location modeled by OPM MEG | Day of the MEG visit (day of inclusion)
  For each patient included, the location of the epileptic focus by MEG OPM will be determined by source modeling applied to the detected epileptic spikes.
  For each patient, the spatial overlap between the area modeled in MEG OPM and the area detected on MRI will be determined, allowing good or poor congruence to be determined.
Proportion of congruence between the location of a hypometabolic focus in FDG PET and the location of epileptic foci modeled by MEG OPM | Day of the MEG visit (day of inclusion)
  For each patient included, the location of the epileptic focus by MEG OPM will be determined by source modeling applied to the detected epileptic spikes.
  For each patient, the spatial overlap between the area modeled by MEG OPM and the area detected by PET-FDG will be determined, allowing good or poor congruence to be determined.
Description of adverse events that occurred and were related to the performance of the MEG OPM examination | From date of inclusion until the end of the study (54 months after inclusion)
  Description of adverse events that occurred and were related to the performance of the MEG OPM examination
Evaluation of patient comfort during OPM MEG recordings using a Likert scale | Day of the MEG visit (day of inclusion)
  Lickert scale with 5 possible responses: very uncomfortable, uncomfortable, neutral, comfortable, very comfortable

CONTACTS AND LOCATIONS:
Overall Officials: Julien JUNG, Professor, Principal Investigator — Hospices Civils de Lyon; Denis SCHWARTZ, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (3):
- France (3):
  - Hôpital Femme-Mère-Enfant, Hospices Civils de Lyon, Service Explorations Fonctionnelles Pédiatriques, Bron
  - Hôpital Neurologique, Hospices Civils de Lyon, Service Explorations Fonctionnelles Neurologiques et Epileptologie, Bron
  - Hôpital de la Timone, AP-HM Service d'Epileptologie et Rythmologie Cérébrale, Marseille